CLINICAL TRIAL: NCT04159532
Title: Comparative Bioavailability Study of Monoglyceride (MAG) Versus Triglyceride (TG) Versus Ethyl Ester (EE) Formulations of Eicosapentaenoic (EPA) and Docosahexaenoic (DHA) Acids. Pilot Study (IO3-03)
Brief Title: Comparative Study of Three Different Formulations of Omega-3 (EPA+DHA)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: SCF Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: IO3-03
Record Dates: First submitted 2019-11-06; First posted 2019-11-12 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Healthy Adults

STUDY DESIGN:
Intervention Model Description: Double-blind, 3-arms parallel randomized study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blinded. Only the sponsor will have access to the randomisation list. No one at the sites will have access to the list.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Monoglyceride (MAG) (Experimental): Group A will receive the omega-3 fatty acids in monoglyceride formulation (MAG). Subjects will receive 1.5g per day of MAG-EPA/MAG-DHA in a proportion of 460:200 for 12 consecutive weeks.
  Interventions: Dietary Supplement: MAG-EPA/MAG-DHA
- Triglyceride (TG) (Active Comparator): Group B will receive the omega-3 fatty acids in triglyceride formulation (TG). Subjects will receive 1.5g per day of TG-EPA/TG-DHA in a proportion of 460:200 for 12 consecutive weeks.
  Interventions: Dietary Supplement: TG-EPA/TG-DHA
- Ethyl Ester(EE) (Active Comparator): Group C will receive the omega-3 fatty acids in Ethyl ester formulation (EE). Subjects will receive 1.5g per day of EE-EPA/EE-DHA in a proportion of 460:200 for 12 consecutive weeks.
  Interventions: Dietary Supplement: EE-EPA/EE-DHA

INTERVENTIONS:
Dietary Supplement: MAG-EPA/MAG-DHA — monoglyceride of eicosapentaenoic acid and docosahexaenoic acid in proportion of 460:200
  Arms: Monoglyceride (MAG)
Dietary Supplement: TG-EPA/TG-DHA — Triglyceride of eicosapentaenoic acid and docosahexaenoic acid in proportion of 460:200
  Arms: Triglyceride (TG)
Dietary Supplement: EE-EPA/EE-DHA — Ethyl ester of eicosapentaenoic acid and docosahexaenoic acid in proportion of 460:200
  Arms: Ethyl Ester(EE)

SUMMARY:
This pilot study aims at comparing the bioavailability of three different formulations of the omega-3 fatty acids eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA). The three formulations are ethyl ester (EE), triglyceride (TG) and monoglyceride (MAG). Thirty six (36) subjects will be divided in three groups of twelve subjects each equally divided in two study sites. Each group will be taking one of the three different formulations of EPA+DHA at a daily dose of 1.5g for a period of 12 weeks. Bioavailability will be measured through omega-3 index (total content of EPA + DHA in red blood cell membranes) at baseline and every four weeks during treatment.

DETAILED DESCRIPTION:
This pilot study aims at comparing the bioavailability of three different formulations of a combination of omega-3 fatty acids eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA) in a standardized proportion of 460:200. The three formulations are ethyl ester (EE), triglyceride (TG) and monoglyceride (MAG) versions of these fatty acids. The formulations are prepared in a way to be similar in proportion of EPA/DHA, in dose and in appearance. Thirty six (36) subjects will be divided in three groups of twelve subjects each, equally divided in two study sites. The study will be randomized and double blinded. Each group will be taking one of the three different formulations of EPA+DHA at a daily dose of 1.5g for a period of 12 weeks. Bioavailability will be measured through omega-3 index (total content of EPA + DHA in red blood cell membranes) at baseline and every four weeks during treatment. After recruitment, subjects will be seen in clinic every four weeks for a total of four (4) study visits during which a blood sample will be taken for analysis of the omega-3 index, the investigational product will be returned and dispensed and finally, adverse events will be noted and followed. Treatment will be self-administered by subjects at home. They will be asked to keep a journal of adverse events, concomitant medication and to note every missed dose as well as significant changes in life habits (smoking, alcohol, sports, food diet and natural health products intake).

ELIGIBILITY:
Inclusion Criteria:

* Participants of at least 19 years of age.
* Availability for the entire duration of the study, willingness to participate as evidenced by the informed consent form duly read and signed by the participant.
* Absence of intellectual problems likely to limit the validity of consent to participate in the study or the compliance with protocol requirements, ability to cooperate adequately, to understand and observe the instructions of the physician or delegates.
* Participant having no difficulty swallowing tablets or capsules.

Exclusion Criteria:

* Known allergy or intolerance to fish or history of allergic reaction attributable to fish or to a compound similar to fish oil.
* Females who are pregnant according to the qualitative pregnancy test or who are lactating.
* Participants who took omega-3 supplements in the previous 60 days before day 1 of the study.
* Difficulty to draw blood by capillary puncture at screening.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-12-18 (Actual); Primary Completion 2021-02-25 (Actual); Study Completion 2021-02-25 (Actual)

PRIMARY OUTCOMES:
Comparing the bioavailability of the three different formulations of omega-3 fatty acids at study. | 12 weeks per subject
  The Omega-3 index (ratio of EPA + DHA content on total fatty acids in red blood cells) will be measured throughout the study (at baseline and every four weeks afterwards) for each subjects. The average value in canadian population is 4.5%, however, for an optimized health, the desired index should be between 8 and 12% of omega-3 in cell membranes. The average omega-3 index curves obtained for each group will be compared to determine which formulation offers the best absorption of omega-3 in the organism.

SECONDARY OUTCOMES:
Incidence of adverse events in subjects treated with EPA +DHA | 16 weeks per subject
  Subjects will be questioned about any changes in their health status throughout the study, and for the 30 days following the end of treatment. All adverse events will recorded and evaluated for severity, causality and expectedness. All serious adverse events will be reported as required.
Compilation of life habits & demographic information | 12 weeks per subject
  Demographic information and life habits will be recorded at screening as to draw a portrait of the subjects baseline status. A follow-up of life habits at every visit will be done afterwards as a way to control any possible bias in outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Fortin, PhD, Principal Investigator — SCF Pharma
Locations (1):
- SCF pharma, Rimouski, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No